CLINICAL TRIAL: NCT01324206
Title: Development of Magnetic Resonance Imaging and Spectroscopy Research Methods for NIA Studies
Brief Title: Development of 3T Magnetic Resonance Research Methods for NIA Studies
Status: Recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080238; 08-AG-0238
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-08

CONDITIONS: Normal Physiology
Keywords: Magnetic Resonance Imaging; Healthy Volunteers; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers, 18 or older years

SUMMARY:
Background:

- Magnetic resonance imaging (MRI) studies provide important information on the structure and function of various body systems, including the brain, muscles, joints, heart, and blood vessels. Scientific applications of MRI scans often use techniques that need to be modified or refined before they are used in clinical studies. To develop and modify these techniques for the new Philips 3T Achieva whole-body MRI scanner, researchers are interested in conducting trial MRI scans on healthy individuals and individuals with conditions that require imaging studies.

Objectives:

- To conduct preliminary trials of the 3T MRI facility to develop and refine MRI scanning procedures.

Eligibility:

- Individuals at least 18 years of age who are able to have magnetic resonance imaging.

Design:

* Participants will be screened with a full medical history and physical examination, as well as blood and urine tests.
* Participants will have an MRI scan using the 3T scanner. Some scans may require the use of a contrast agent or radiotracer, which is a small amount of radioactive substance that will be injected before the start of the scan. Some participants may be asked to perform tasks of thinking and movement while in the scanner, in order to test the procedures required for a functional MRI scan.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
Study Description:

The purpose of this protocol is to permit use of the magnetic resonance imaging (MRI) facility for the development and refinement of MRI and spectroscopy (MRIS) scanning procedures. The information obtained through these methodological assessments will be essential future clinical research investigations conducted through the NIA under specific protocols. Additionally, this data can be utilized in already approved NIA studies for comparison purposes.

Objectives:

Primary Objective: To develop and refine specific MR imaging and spectroscopy methods.

Secondary Objectives: To allow pilot tests of procedures for development and refinement of motor or cognitive activation paradigms.

Endpoints:

Development of noninvasive MR biomarkers to assess longevity, healthy longevity, physical disability, cognitive impairment, and frailty.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

* Ability of subject to understand the study and stated willingness to comply with all study procedures.
* Male or female, age > 18years.
* Able to speak and read English.
* Capable of providing informed consent.
* Subjects or persons identified by an investigator to have a condition of interest for exploratory studies as it relates to aging. These participants are not being scanned for diagnostic purposes.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Has condition and/or non-removable device contraindicated for MRI as per the MRI eligibility form.
* Weight > 300lbs (MRI scanner weight limit)
* Is currently pregnant or a nursing mother.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, male and female, 18yrs and older
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-11-03 (Actual)

PRIMARY OUTCOMES:
Develop and refine scanning procedures | 2 months
  To develop and refine specific imaging and spectroscopic methods.

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha Bouhrara, Ph.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is ongoing discussion within the NIA IRP and a plan has not been finalized yet.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-AG-0238.html